CLINICAL TRIAL: NCT02091271
Title: Screening Protocol to Evaluate Volunteers for NIA Approved Studies
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903335; 03-AG-N335
Record Dates: First submitted 2013-09-20; First posted 2014-03-19 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Volunteers
Keywords: Evaluation; Research; Healthy Volunteers

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The National Institute on Aging (NIA) Intramural Research Program (IRP) has a number ofiRB approved research studies involving human subjects, both normal volunteers and patients. As a means of identifying interested volunteers and other participants in the research process, this screening mechanism is established to identif'y potential eligible participants for NlA protocols.

To participate, volunteers/patients must meet the specific requirements of at least one of the available NlA research studies; this protocol serves as a first step for admitting volunteers/patients to an appropriate approved protocol and creating a contact database for approved NlA studies.

This protocol will facilitate their recruitment into NIA approved studies and provide NlA staff the opportunity to examine subjects where diagnostic observations can be documented and evaluated for research potential.

DETAILED DESCRIPTION:
The screening protocol is designed to evaluate volunteers/patients for participation in IRB approved clinical studies of the National Institute on Aging (NIA). An additional purpose of this protocol is to develop a registry of individuals who have been evaluated through the NIA Clinical Research Unit screening clinic. To participate, volunteers/patients must meet the specific requirements of at least one of the available NIA research studies. This protocol serves as a first step for admitting volunteers/patients to an appropriate approved protocol, and it is used to develop a registry of individuals who meet eligibility criteria for existing research projects.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. All volunteers/patients who meet the criteria of an approved NIA protocol.
  2. People with diagnosed or undiagnosed conditions
  3. Patients may be eligible if they have rare, unusual, interesting or unknown conditions that require diagnosis

EXCLUSION CRITERIA:

1. Subjects unable to provide informed consent.
2. The volunteer/patient does not meet the criteria of any approved NIA protocol and does not wish to remain in the contact database for future studies.
3. Volunteer/patient has contacted the NIA Clinical Research Protocol Office and notified them that they would like to be removed and no longer contacted for NIA approved studies. They will be removed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2003-02-28 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Develop a registry of individuals who meet eligibility criteria forexisting research projects | ongoing
Evaluate volunteers/patients for participation in IRB approved clinicalstudies at NIA | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Chee W Chia, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States